CLINICAL TRIAL: NCT03279198
Title: Increasing Colorectal and Breast Cancer Screening in Women
Acronym: COBRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Victoria L. Champion, Distinguished Professor Edward and Sara Stam Culliper named Professor Associate Director Cancer Prevention and Control, Indiana University
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 1009001808; 5R01CA136940-05 (NIH)
Record Dates: First submitted 2017-08-22; First posted 2017-09-12 (Actual); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer Female; Colorectal Cancer
Keywords: breast cancer screening; colorectal cancer screening; cervical cancer screening; cancer screening beliefs; cost-effectiveness; demographics; tailored intervention
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: We propose a prospective randomized 2x2 factorial design: 1)usual care; 2) a TIWeb; 3) a Cancer Screening Call (CSC), and 4 a TIWEB+ a Cancer Screening Call (CSC). The intervention will be tested in 2 groups of women. Group A will include women who are nonadherent to CRC but adherent to BC screening guidelines. Group B will include women who are nonadherent to both CRC and BC screening guidelines.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual Care (UC) (Placebo Comparator): The usual care group received usual care that varies dependent upon the practice setting.
  Interventions: Behavioral: UC
- TIWeb (Active Comparator): TIWeb (Tailored Web Intervention) program is interactive and tailored to the participant's individual beliefs and demographics. Individuals receiving the TIWeb will be given information that allows them to call and receive an FOBT kit in the mail or schedule an appropriate CRC test and/or mammogram.
  Interventions: Behavioral: TIWeb
- Cancer Screening Call (CSC) (Active Comparator): CSC - a telephone counseling call during which the participant is given the opportunity to complete CRC screening (FOBT or a colonoscopy) and/or mammography screening.The CSC included tailored counseling as well as the ability to schedule BC and CRC screening tests.
  Interventions: Behavioral: CSC
- TIWeb+CSC (Active Comparator): TIWeb + CSC ((Tailored web intervetion+Cancer screening) group receive a mailed TIWeb, which is followed in four weeks by a CSC with the same opportunity to receive FOBT kits or schedule a colonoscopy and/or mammogram. The nurse counselor, knowing the participant is a good candidate for screening tests, will be trained to schedule CRC or BC screening appointments or to mail FOBT kits to individuals in the intervention groups even if they have not had a recent clinic visit.
  Interventions: Behavioral: TIWeb+CSC

INTERVENTIONS:
Behavioral: TIWeb — Intervention: TIWeb program is interactive and tailored to the participant's individual beliefs and demographics. Individuals receiving the TIWeb will be given information that allows them to call and receive an FOBT kit in the mail or schedule an appropriate CRC test and/or mammogram.
  Other Names: Tailored Web Intervention
  Arms: TIWeb
Behavioral: CSC — Intervention: CSC - a telephone counseling call during which the participant is given the opportunity to complete CRC screening (FOBT or a colonoscopy) and/or mammography screening.The CSC included tailored counseling as well as the ability to schedule BC and CRC screening tests.
  Other Names: Cancer Screening Call
  Arms: Cancer Screening Call (CSC)
Behavioral: UC — Intervention: The usual care group received usual care that varies dependent upon the practice setting.
  Other Names: Usual Care
  Arms: Usual Care (UC)
Behavioral: TIWeb+CSC — Intervention: TIWeb + CSC ((Tailored web intervetion+Cancer screening) group receive a mailed TIWeb, which is followed in four weeks by a CSC with the same opportunity to receive FOBT kits or schedule a colonoscopy and/or mammogram. The nurse counselor, knowing the participant is a good candidate for screening tests, will be trained to schedule CRC or BC screening appointments or to mail FOBT kits to individuals in the intervention groups even if they have not had a recent clinic visit.
  Other Names: Tailored Web Intervention + Cancer Screening Call
  Arms: TIWeb+CSC

SUMMARY:
This study compares the efficacy (adherence and stage) of four interventions to promote colorectal (CRC) and breast cancer (BC) screenings among women ages 50 to 75. They are:

1. usual care;
2. a TIWeb (tailored intervention Website)
3. a CSC (cancer screening call) and
4. TIWeb + a CSC. This study also compares the cost-effectiveness of the 4 interventions to promote CRC and BC screening among women ages 50 to 75.

DETAILED DESCRIPTION:
This study addresses innovative approaches to increase adherence to screening tests for colorectal and breast cancer - two cancers that have the greatest impact on female cancer mortality in the United States.The cancer burden in women could be significantly reduced by increasing participation in recommended screening for colorectal cancer (CRC) and breast cancer (BC) in all eligible women. This research tests intervention to simultaneously increase both CRC and BC screening using behavior change strategies, and also estimates the efficacy and cost-effectiveness of the interventions. Two groups of women, Group A (adherent to BC screening guidelines, but NOT to CRC screening guidelines) and Group B (non-adherent to BC & CRC guidelines) are randomized to 1. Usual Care, 2. TIWeb, 3. CSC and 4. TIWeb +CSC.

ELIGIBILITY:
Inclusion Criteria:

* a patient of any of the participating physicians
* not having had a fecal occult blood test (fobt) in the last 12 months
* not having had a fecal immunochemical test (fit) in the past 15 months
* not having had sigmoidoscopy more than 5 years ago
* not having had a colonoscopy more than 10 years ago
* have high-speed internet access

Exclusion Criteria

* a personal history of colorectal cancer
* a personal history of breast cancer
* a personal history of colorectal polyps
* a personal history of inflammatory bowel disease
* having any medical conditions that would prohibit a mammogram or CRC screening
* have already had CRC screening

Ages: 50 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Women between the ages from 50 - 75.
Enrollment: 1196 (Actual)
Dates: Start 2010-07-22 (Actual); Primary Completion 2015-09-15 (Actual); Study Completion 2017-05-31 (Actual)

PRIMARY OUTCOMES:
Primary Outcome -differences in CRC screening adherence, when controlling for adherence to BC screening at baseline, among women who are randomized to 1) usual care; 2) a TIWeb; 3) a CSC, and 4) a TIWeb plus a CSC. | 6 months from the baseline measure
  any CRC test (either a stool test or colonoscopy) receipt of a stool test or a colonoscopy
Primary Outcome:differences in stage of adoption (precontemplation, contemplation, action) when controlling for adherence to BC screening at baseline, among women who are randomized to 1) usual care; 2) a TIWeb; 3) a CSC, and 4) a TIWeb plus a CSC. | 6 months from the baseline measure
  Forward stage movement is the desired outcome -determining any forward stage movement in considering CRC screening either from Precontemplation to contemplation or from precontemplation to action

SECONDARY OUTCOMES:
Secondary outcome:Intervention Costs | 6 months from the baseline measure
  Comparing the cost-effectiveness of four conditions to promote CRC and BC screening , there will be differences in adherence to both CRC and BC screening and stage of adoption, among women who are randomized to 1) usual care; 2) a TIWeb; 3) a CSC, and 4) a TIWeb plus a CSC.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Champion, PhD, Principal Investigator — Indiana University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
De-identified IPD will be made available to other researchers through a HIPAA compliant data storage system (Box Health) that is password protected.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: January 1st, 2017 - March 31st, 2020.
Access Criteria: Research staff solely associated with the study and/or Graduate or Post-Doc students-who are writing related manuscripts - who have been given permission by the Principal Investigator, Victoria Champion can submit a request.

REFERENCES:
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] Smith RA, Cokkinides V, Eyre HJ. American Cancer Society guidelines for the early detection of cancer, 2006. CA Cancer J Clin. 2006 Jan-Feb;56(1):11-25; quiz 49-50. doi: 10.3322/canjclin.56.1.11. PMID 16449183
- [Background] American Cancer Society. Report finds historic drop in total number of cancer deaths. 2006 [updated 2006; cited]; Available from: http://www.cancer.org/docroot/MED/content/MED_2_lx_American_Cancer_Society_Report_Finds_Drop _in_Total_Cancer_Deaths.asp
- [Background] Breen N, A Cronin K, Meissner HI, Taplin SH, Tangka FK, Tiro JA, McNeel TS. Reported drop in mammography : is this cause for concern? Cancer. 2007 Jun 15;109(12):2405-9. doi: 10.1002/cncr.22723. PMID 17503429
- [Background] Prochaska JJ, Spring B, Nigg CR. Multiple health behavior change research: an introduction and overview. Prev Med. 2008 Mar;46(3):181-8. doi: 10.1016/j.ypmed.2008.02.001. Epub 2008 Feb 6. PMID 18319098
- [Background] Stockwell DH, Woo P, Jacobson BC, Remily R, Syngal S, Wolf J, Farraye FA. Determinants of colorectal cancer screening in women undergoing mammography. Am J Gastroenterol. 2003 Aug;98(8):1875-80. doi: 10.1111/j.1572-0241.2003.07577.x. PMID 12907347
- [Background] Solomon D, Breen N, McNeel T. Cervical cancer screening rates in the United States and the potential impact of implementation of screening guidelines. CA Cancer J Clin. 2007 Mar-Apr;57(2):105-11. doi: 10.3322/canjclin.57.2.105. PMID 17392387
- [Background] Katz ML, Tatum CM, Degraffinreid CR, Dickinson S, Paskett ED. Do cervical cancer screening rates increase in association with an intervention designed to increase mammography usage? J Womens Health (Larchmt). 2007 Jan-Feb;16(1):24-35. doi: 10.1089/jwh.2006.0071. PMID 17324094
- [Background] Champion VL. Strategies to increase mammography utilization. Med Care. 1994 Feb;32(2):118-29. doi: 10.1097/00005650-199402000-00003. PMID 8302104
- [Background] Skinner CS, Strecher VJ, Hospers H. Physicians' recommendations for mammography: do tailored messages make a difference? Am J Public Health. 1994 Jan;84(1):43-9. doi: 10.2105/ajph.84.1.43. PMID 8279610
- [Background] Taplin SH, Barlow WE, Ludman E, MacLehos R, Meyer DM, Seger D, Herta D, Chin C, Curry S. Testing reminder and motivational telephone calls to increase screening mammography: a randomized study. J Natl Cancer Inst. 2000 Feb 2;92(3):233-42. doi: 10.1093/jnci/92.3.233. PMID 10655440
- [Background] American Cancer Society. Cancer Facts & Figures 2009. Atlanta; 2009 Contract No.: Document Number|.
- [Background] Shapiro JA, Seeff LC, Nadel MR. Colorectal cancer-screening tests and associated health behaviors. Am J Prev Med. 2001 Aug;21(2):132-7. doi: 10.1016/s0749-3797(01)00329-4. PMID 11457633
- [Background] Saywell RM Jr, Champion VL, Skinner CS, McQuillen D, Martin D, Maraj M. Cost-effectiveness comparison of five interventions to increase mammography screening. Prev Med. 1999 Nov;29(5):374-82. doi: 10.1006/pmed.1999.0568. PMID 10564629
- [Background] Saywell RM Jr, Champion VL, Zollinger TW, Maraj M, Skinner CS, Zoppi KA, Muegge CM. The cost effectiveness of 5 interventions to increase mammography adherence in a managed care population. Am J Manag Care. 2003 Jan;9(1):33-44. PMID 12549813
- [Background] Noar SM, Chabot M, Zimmerman RS. Applying health behavior theory to multiple behavior change: considerations and approaches. Prev Med. 2008 Mar;46(3):275-80. doi: 10.1016/j.ypmed.2007.08.001. Epub 2007 Aug 11. PMID 17825898
- [Background] Champion V, Springston J, Hui S, Saywell RM, Jr., Zollinger TW, Ray D. Community intervention to increase mammography screening (funded research R01CA77736). Bethesda, MD: National Cancer Institute; 1998-2002 Contract No.: Document Number|.
- [Background] American Cancer Society. Cancer prevention & early detection facts & figures 2005. Atlanta: American Cancer Society; 2005 Contract No.: Document Number|.
- [Background] Mandel JS, Bond JH, Church TR, Snover DC, Bradley GM, Schuman LM, Ederer F. Reducing mortality from colorectal cancer by screening for fecal occult blood. Minnesota Colon Cancer Control Study. N Engl J Med. 1993 May 13;328(19):1365-71. doi: 10.1056/NEJM199305133281901. PMID 8474513
- [Background] Winawer SJ, Fletcher RH, Miller L, Godlee F, Stolar MH, Mulrow CD, Woolf SH, Glick SN, Ganiats TG, Bond JH, Rosen L, Zapka JG, Olsen SJ, Giardiello FM, Sisk JE, Van Antwerp R, Brown-Davis C, Marciniak DA, Mayer RJ. Colorectal cancer screening: clinical guidelines and rationale. Gastroenterology. 1997 Feb;112(2):594-642. doi: 10.1053/gast.1997.v112.agast970594. No abstract available. PMID 9024315
- [Background] Shapiro S. Periodic screening for breast cancer: the HIP Randomized Controlled Trial. Health Insurance Plan. J Natl Cancer Inst Monogr. 1997;(22):27-30. doi: 10.1093/jncimono/1997.22.27. PMID 9709271
- [Background] Tabar L, Fagerberg CJ, Gad A, Baldetorp L, Holmberg LH, Grontoft O, Ljungquist U, Lundstrom B, Manson JC, Eklund G, et al. Reduction in mortality from breast cancer after mass screening with mammography. Randomised trial from the Breast Cancer Screening Working Group of the Swedish National Board of Health and Welfare. Lancet. 1985 Apr 13;1(8433):829-32. doi: 10.1016/s0140-6736(85)92204-4. PMID 2858707
- [Background] Tabar L, Fagerberg G, Duffy SW, Day NE, Gad A, Grontoft O. Update of the Swedish two-county program of mammographic screening for breast cancer. Radiol Clin North Am. 1992 Jan;30(1):187-210. PMID 1732926
- [Background] Tabar L, Faberberg G, Day NE, Holmberg L. What is the optimum interval between mammographic screening examinations? An analysis based on the latest results of the Swedish two-county breast cancer screening trial. Br J Cancer. 1987 May;55(5):547-51. doi: 10.1038/bjc.1987.112. PMID 3606947
- [Background] Nystrom L, Rutqvist LE, Wall S, Lindgren A, Lindqvist M, Ryden S, Andersson I, Bjurstam N, Fagerberg G, Frisell J, et al. Breast cancer screening with mammography: overview of Swedish randomised trials. Lancet. 1993 Apr 17;341(8851):973-8. doi: 10.1016/0140-6736(93)91067-v. PMID 8096941
- [Background] Andersson I, Aspegren K, Janzon L, Landberg T, Lindholm K, Linell F, Ljungberg O, Ranstam J, Sigfusson B. Mammographic screening and mortality from breast cancer: the Malmo mammographic screening trial. BMJ. 1988 Oct 15;297(6654):943-8. doi: 10.1136/bmj.297.6654.943. PMID 3142562
- [Background] Frisell J, Eklund G, Hellstrom L, Lidbrink E, Rutqvist LE, Somell A. Randomized study of mammography screening--preliminary report on mortality in the Stockholm trial. Breast Cancer Res Treat. 1991 Mar;18(1):49-56. doi: 10.1007/BF01975443. PMID 1854979
- [Background] Roberts MM, Alexander FE, Anderson TJ, Chetty U, Donnan PT, Forrest P, Hepburn W, Huggins A, Kirkpatrick AE, Lamb J, et al. Edinburgh trial of screening for breast cancer: mortality at seven years. Lancet. 1990 Feb 3;335(8684):241-6. doi: 10.1016/0140-6736(90)90066-e. PMID 1967717
- [Background] Miller AB, Howe GR, Wall C. The National Study of Breast Cancer Screening Protocol for a Canadian Randomized Controlled trial of screening for breast cancer in women. Clin Invest Med. 1981;4(3-4):227-58. No abstract available. PMID 6802546
- [Background] Miller AB, Baines CJ, To T, Wall C. Canadian National Breast Screening Study: 1. Breast cancer detection and death rates among women aged 40 to 49 years. CMAJ. 1992 Nov 15;147(10):1459-76. PMID 1423087
- [Background] Miller AB, Baines CJ, To T, Wall C. Canadian National Breast Screening Study: 2. Breast cancer detection and death rates among women aged 50 to 59 years. CMAJ. 1992 Nov 15;147(10):1477-88. PMID 1423088
- [Background] Agency for Healthcare Research and Quality. Screening for breast cancer. Recommendations and rationale: Agency for Healthcare Research and Quality; 2002 February 2002 Contract No.: Document Number|.
- [Background] Quigley TF, Davis RH Jr, Larson LW, Leger MM, McNellis R, Muma RD, Toth SA. Making decisions on breast cancer screening. JAAPA. 2002 Jul;15(7):11-3. No abstract available. PMID 12192828
- [Background] Smith RA, Cokkinides V, Brawley OW. Cancer screening in the United States, 2008: a review of current American Cancer Society guidelines and cancer screening issues. CA Cancer J Clin. 2008 May-Jun;58(3):161-79. doi: 10.3322/CA.2007.0017. Epub 2008 Apr 28. PMID 18443206
- [Background] Kreuter M, Lezin N, Krueter M, Green L. Community health promotion ideas that work. Boston: Jones and Bartlet; 1998.
- [Background] Goldstein MG, Whitlock EP, DePue J; Planning Committee of the Addressing Multiple Behavioral Risk Factors in Primary Care Project. Multiple behavioral risk factor interventions in primary care. Summary of research evidence. Am J Prev Med. 2004 Aug;27(2 Suppl):61-79. doi: 10.1016/j.amepre.2004.04.023. PMID 15275675
- [Background] Beeker C, Kraft JM, Southwell BG, Jorgensen CM. Colorectal cancer screening in older men and women: qualitative research findings and implications for intervention. J Community Health. 2000 Jun;25(3):263-78. doi: 10.1023/a:1005104406934. PMID 10868818
- [Background] Price JH, Colvin TL, Smith D. Prostate cancer: perceptions of African-American males. J Natl Med Assoc. 1993 Dec;85(12):941-7. PMID 8126745
- [Background] Myers RE, Trock BJ, Lerman C, Wolf T, Ross E, Engstrom PF. Adherence to colorectal cancer screening in an HMO population. Prev Med. 1990 Sep;19(5):502-14. doi: 10.1016/0091-7435(90)90049-p. PMID 2235919
- [Background] Farrands PA, Hardcastle JD, Chamberlain J, Moss S. Factors affecting compliance with screening for colorectal cancer. Community Med. 1984 Feb;6(1):12-9. No abstract available. PMID 6705494
- [Background] Brown ML, Potosky AL, Thompson GB, Kessler LG. The knowledge and use of screening tests for colorectal and prostate cancer: data from the 1987 National Health Interview Survey. Prev Med. 1990 Sep;19(5):562-74. doi: 10.1016/0091-7435(90)90054-n. PMID 2235923
- [Background] Manne S, Markowitz A, Winawer S, Meropol NJ, Haller D, Rakowski W, Babb J, Jandorf L. Correlates of colorectal cancer screening compliance and stage of adoption among siblings of individuals with early onset colorectal cancer. Health Psychol. 2002 Jan;21(1):3-15. PMID 11846342
- [Background] Myers RE, Ross E, Jepson C, Wolf T, Balshem A, Millner L, Leventhal H. Modeling adherence to colorectal cancer screening. Prev Med. 1994 Mar;23(2):142-51. doi: 10.1006/pmed.1994.1020. PMID 8047519
- [Background] Polednak AP. Knowledge of colorectal cancer and use of screening tests in persons 40-74 years of age. Prev Med. 1990 Mar;19(2):213-26. doi: 10.1016/0091-7435(90)90022-c. PMID 2359743
- [Background] Manne S, Markowitz A, Winawer S, Guillem J, Meropol NJ, Haller D, Jandorf L, Rakowski W, Babb J, Duncan T. Understanding intention to undergo colonoscopy among intermediate-risk siblings of colorectal cancer patients: a test of a mediational model. Prev Med. 2003 Jan;36(1):71-84. doi: 10.1006/pmed.2002.1122. PMID 12473427
- [Background] Rawl SM, Menon U, Champion VL, May FE, Loehrer P Sr, Hunter C, Azzouz F, Monahan PO, Skinner CS. Do benefits and barriers differ by stage of adoption for colorectal cancer screening? Health Educ Res. 2005 Apr;20(2):137-48. doi: 10.1093/her/cyg110. Epub 2004 Aug 16. PMID 15314036
- [Background] Prochaska JO, Velicer WF. The transtheoretical model of health behavior change. Am J Health Promot. 1997 Sep-Oct;12(1):38-48. doi: 10.4278/0890-1171-12.1.38. PMID 10170434
- [Background] Champion VL, Skinner CS. Differences in perceptions of risk, benefits, and barriers by stage of mammography adoption. J Womens Health (Larchmt). 2003 Apr;12(3):277-86. doi: 10.1089/154099903321667618. PMID 12804358
- [Background] Madlensky L, Esplen MJ, Gallinger S, McLaughlin JR, Goel V. Relatives of colorectal cancer patients: factors associated with screening behavior. Am J Prev Med. 2003 Oct;25(3):187-94. doi: 10.1016/s0749-3797(03)00202-2. PMID 14507524
- [Background] Hay JL, Buckley TR, Ostroff JS. The role of cancer worry in cancer screening: a theoretical and empirical review of the literature. Psychooncology. 2005 Jul;14(7):517-34. doi: 10.1002/pon.864. PMID 15490428
- [Background] Andersen MR, Smith R, Meischke H, Bowen D, Urban N. Breast cancer worry and mammography use by women with and without a family history in a population-based sample. Cancer Epidemiol Biomarkers Prev. 2003 Apr;12(4):314-20. PMID 12692105
- [Background] Skinner CS, Champion VL, Menon U, Seshadri R. Racial and educational differences in mammography-related perceptions among 1,336 nonadherent women. Journal of Psychosocial Oncology. 2002;20:1-18.
- [Background] Lauver DR, Henriques JB, Settersten L, Bumann MC. Psychosocial variables, external barriers, and stage of mammography adoption. Health Psychol. 2003 Nov;22(6):649-53. doi: 10.1037/0278-6133.22.6.649. PMID 14640864
- [Background] Taylor R, Ivanov O, Page A, Brotherton J, Achat H, Close G. Predictors of non-attendance from BreastScreen NSW in women who report current mammography screening. Aust N Z J Public Health. 2003 Dec;27(6):581-7. doi: 10.1111/j.1467-842x.2003.tb00603.x. PMID 14723404
- [Background] Friedman LC, Webb JA, Richards CS, Plon SE. Psychological and behavioral factors associated with colorectal cancer screening among Ashkenazim. Prev Med. 1999 Aug;29(2):119-25. doi: 10.1006/pmed.1999.0508. PMID 10446038
- [Background] Gordon NP, Rundall TG, Parker L. Type of health care coverage and the likelihood of being screened for cancer. Med Care. 1998 May;36(5):636-45. doi: 10.1097/00005650-199805000-00004. PMID 9596055
- [Background] Holt WS Jr. Factors affecting compliance with screening sigmoidoscopy. J Fam Pract. 1991 Jun;32(6):585-9. PMID 2040883
- [Background] Leard LE, Savides TJ, Ganiats TG. Patient preferences for colorectal cancer screening. J Fam Pract. 1997 Sep;45(3):211-8. PMID 9300000
- [Background] Lewis SF, Jensen NM. Screening sigmoidoscopy. Factors associated with utilization. J Gen Intern Med. 1996 Sep;11(9):542-4. doi: 10.1007/BF02599602. PMID 8905504
- [Background] McCarthy BD, Moskowitz MA. Screening flexible sigmoidoscopy: patient attitudes and compliance. J Gen Intern Med. 1993 Mar;8(3):120-5. doi: 10.1007/BF02599753. PMID 8455106
- [Background] Rawl SM, Menon U, Champion VL, Foster JL, Skinner CS. Colorectal cancer screening beliefs. Focus groups with first-degree relatives. Cancer Pract. 2000 Jan-Feb;8(1):32-7. doi: 10.1046/j.1523-5394.2000.81006.x. PMID 10732537
- [Background] Lipkus IM, Rimer BK, Halabi S, Strigo TS. Can tailored interventions increase mammography use among HMO women? Am J Prev Med. 2000 Jan;18(1):1-10. doi: 10.1016/s0749-3797(99)00106-3. PMID 10808977
- [Background] Rakowski W, Ehrich B, Goldstein MG, Rimer BK, Pearlman DN, Clark MA, Velicer WF, Woolverton H 3rd. Increasing mammography among women aged 40-74 by use of a stage-matched, tailored intervention. Prev Med. 1998 Sep-Oct;27(5 Pt 1):748-56. doi: 10.1006/pmed.1998.0354. PMID 9808807
- [Background] Noar SM, Benac CN, Harris MS. Does tailoring matter? Meta-analytic review of tailored print health behavior change interventions. Psychol Bull. 2007 Jul;133(4):673-93. doi: 10.1037/0033-2909.133.4.673. PMID 17592961
- [Background] King ES, Rimer BK, Seay J, Balshem A, Engstrom PF. Promoting mammography use through progressive interventions: is it effective? Am J Public Health. 1994 Jan;84(1):104-6. doi: 10.2105/ajph.84.1.104. PMID 8279593
- [Background] Marcus AC, Bastani R, Reardon K, Karlins S, Das IP, Van Herle MP, McClatchey MW, Crane LA. Proactive screening mammography counseling within the Cancer Information Service: results from a randomized trial. J Natl Cancer Inst Monogr. 1993;(14):119-29. PMID 8123349
- [Background] Rimer BK, Halabi S, Sugg Skinner C, Lipkus IM, Strigo TS, Kaplan EB, Samsa GP. Effects of a mammography decision-making intervention at 12 and 24 months. Am J Prev Med. 2002 May;22(4):247-57. doi: 10.1016/s0749-3797(02)00417-8. PMID 11988381
- [Background] Champion VL, Skinner CS, Menon U, Seshadri R, Anzalone DC, Rawl SM. Comparisons of tailored mammography interventions at two months postintervention. Ann Behav Med. 2002 Summer;24(3):211-8. doi: 10.1207/S15324796ABM2403_06. PMID 12173678
- [Background] Kreuter MW, Farrell D, Olevitch L, Brennan L. Tailoring health messages: customizing communication with computer technology. Mahwah: Lawrence Erlbaum Associates; 2000.
- [Background] Champion VL, Springston JK, Zollinger TW, Saywell RM Jr, Monahan PO, Zhao Q, Russell KM. Comparison of three interventions to increase mammography screening in low income African American women. Cancer Detect Prev. 2006;30(6):535-44. doi: 10.1016/j.cdp.2006.10.003. Epub 2006 Nov 15. PMID 17110056
- [Background] Skinner CS, Kobrin SC, Monahan PO, Daggy J, Menon U, Todora HS, Champion VL. Tailored interventions for screening mammography among a sample of initially non-adherent women: when is a booster dose important? Patient Educ Couns. 2007 Jan;65(1):87-94. doi: 10.1016/j.pec.2006.06.013. Epub 2006 Jul 26. PMID 16872787
- [Background] Strecher VJ, Kreuter M, Den Boer DJ, Kobrin S, Hospers HJ, Skinner CS. The effects of computer-tailored smoking cessation messages in family practice settings. J Fam Pract. 1994 Sep;39(3):262-70. PMID 8077905
- [Background] Skinner CS, Campbell MK, Rimer BK, Curry S, Prochaska JO. How effective is tailored print communication? Ann Behav Med. 1999 Fall;21(4):290-8. doi: 10.1007/BF02895960. PMID 10721435
- [Background] Clark MA, Rakowski W, Ehrich B, Rimer BK, Velicer WF, Dube CE, Pearlman DN, Peterson KK, Goldstein M. The effect of a stage-matched and tailored intervention on repeat mammography(1). Am J Prev Med. 2002 Jan;22(1):1-7. doi: 10.1016/s0749-3797(01)00406-8. PMID 11777672
- [Background] Jerant A, Kravitz RL, Rooney M, Amerson S, Kreuter M, Franks P. Effects of a tailored interactive multimedia computer program on determinants of colorectal cancer screening: a randomized controlled pilot study in physician offices. Patient Educ Couns. 2007 Apr;66(1):67-74. doi: 10.1016/j.pec.2006.10.009. Epub 2006 Dec 6. PMID 17156968
- [Background] Powe BD, Weinrich S. An intervention to decrease cancer fatalism among rural elders. Oncol Nurs Forum. 1999 Apr;26(3):583-8. PMID 10214599
- [Background] Powe BD. Promoting fecal occult blood testing in rural African American women. Cancer Pract. 2002 May-Jun;10(3):139-46. doi: 10.1046/j.1523-5394.2002.103008.x. PMID 11972568
- [Background] Tilley BC, Vernon SW, Myers R, Glanz K, Lu M, Hirst K, Kristal AR. The Next Step Trial: impact of a worksite colorectal cancer screening promotion program. Prev Med. 1999 Mar;28(3):276-83. doi: 10.1006/pmed.1998.0427. PMID 10072746
- [Background] Pignone M, Harris R, Kinsinger L. Videotape-based decision aid for colon cancer screening. A randomized, controlled trial. Ann Intern Med. 2000 Nov 21;133(10):761-9. doi: 10.7326/0003-4819-133-10-200011210-00008. PMID 11085838
- [Background] Wardle J, Williamson S, McCaffery K, Sutton S, Taylor T, Edwards R, Atkin W. Increasing attendance at colorectal cancer screening: testing the efficacy of a mailed, psychoeducational intervention in a community sample of older adults. Health Psychol. 2003 Jan;22(1):99-105. doi: 10.1037//0278-6133.22.1.99. PMID 12558207
- [Background] Rimal RN, Flora JA. Interactive technology attributes in health promotion: practical and theoretical issues. In: Street RL, Gold WR, Manning T, editors. Health Promotion and Interactive Technology: Theoretical Applications and Future Directions. Mahwah: Lawrence Erlbaum Associates; 1997. p. 19- 38.
- [Background] Ellis LB. Computer-based patient education. Prim Care. 1985 Sep;12(3):547-55. PMID 3906726
- [Background] Ellis LB, Raines JR. Health education using microcomputers: initial acceptability. Prev Med. 1981 Jan;10(1):77-84. doi: 10.1016/0091-7435(81)90008-6. No abstract available. PMID 7015306
- [Background] Vargo G. Computer assisted patient education in the ambulatory care setting. Comput Nurs. 1991 Sep-Oct;9(5):168-9. No abstract available. PMID 1933657
- [Background] Luker KA, Box D. The response of nurses towards the management and teaching of patients on continuous ambulatory peritoneal dialysis (CAPD). Int J Nurs Stud. 1986;23(1):51-9. doi: 10.1016/0020-7489(86)90037-4. PMID 3632951
- [Background] Pingree S, Hawkins RP, Gustafson DH, Boberg E, Bricker E, Wise M, et al. Will the disadvantaged ride the information highway? Hopeful answers from a computer-based health crisis system. Journal of Broadcasting & Electronic Media. 1996;40(3):331-53.
- [Background] Lewis D. Computer-based approaches to patient education: a review of the literature. J Am Med Inform Assoc. 1999 Jul-Aug;6(4):272-82. doi: 10.1136/jamia.1999.0060272. PMID 10428001
- [Background] Tamm EP, Raval BK, Huynh PT. Evaluation of the quality of self-education mammography material available for patients on the Internet. Acad Radiol. 2000 Mar;7(3):137-41. doi: 10.1016/s1076-6332(00)80113-0. PMID 10730807
- [Background] Shaw MJ, Beebe TJ, Tomshine PA, Adlis SA, Cass OW. A randomized, controlled trial of interactive, multimedia software for patient colonoscopy education. J Clin Gastroenterol. 2001 Feb;32(2):142-7. doi: 10.1097/00004836-200102000-00010. PMID 11205650
- [Background] CDRinfo.com. Blu-ray penetration on Rise, Report Says2008 [cited 2008 October 20]: Available from: http://www.cdrinfo.com/sections/news/Details.aspx?NewsId=22933.
- [Background] Nielsen. Neilsen Media Report. 2008 [updated 2008; cited 2008 September 15]; Available from: htpp://www.nielsenmedia.com.
- [Background] Sarfaty M, Wender R. How to increase colorectal cancer screening rates in practice. CA Cancer J Clin. 2007 Nov-Dec;57(6):354-66. doi: 10.3322/CA.57.6.354. PMID 17989130
- [Background] Stone EG, Morton SC, Hulscher ME, Maglione MA, Roth EA, Grimshaw JM, Mittman BS, Rubenstein LV, Rubenstein LZ, Shekelle PG. Interventions that increase use of adult immunization and cancer screening services: a meta-analysis. Ann Intern Med. 2002 May 7;136(9):641-51. doi: 10.7326/0003-4819-136-9-200205070-00006. PMID 11992299
- [Background] Castro CM, King AC. Telephone-assisted counseling for physical activity. Exerc Sport Sci Rev. 2002 Apr;30(2):64-8. doi: 10.1097/00003677-200204000-00004. PMID 11991539
- [Background] Fox SA, Klos DS, Worthen NJ, Pennington E, Bassett LW, Gold RH. Improving the adherence of urban women to mammography guidelines: strategies for radiologists. Radiology. 1990 Jan;174(1):203-6. doi: 10.1148/radiology.174.1.2294548.
- [Background] Frazier AL, Colditz GA, Fuchs CS, Kuntz KM. Cost-effectiveness of screening for colorectal cancer in the general population. JAMA. 2000 Oct 18;284(15):1954-61. doi: 10.1001/jama.284.15.1954. PMID 11035892
- [Background] Pignone M, Saha S, Hoerger T, Mandelblatt J. Cost-effectiveness analyses of colorectal cancer screening: a systematic review for the U.S. Preventive Services Task Force. Ann Intern Med. 2002 Jul 16;137(2):96-104. doi: 10.7326/0003-4819-137-2-200207160-00007. PMID 12118964
- [Background] Andersen MR, Urban N, Ramsey S, Briss PA. Examining the cost-effectiveness of cancer screening promotion. Cancer. 2004 Sep 1;101(5 Suppl):1229-38. doi: 10.1002/cncr.20511. PMID 15316909
- [Background] Abrams DB, Mills S, Bulger D. Challenges and future directions for tailored communication research. Ann Behav Med. 1999 Fall;21(4):299-306. doi: 10.1007/BF02895961. PMID 10721436
- [Background] Emmons KM, McBride CM, Puleo E, Pollak KI, Marcus BH, Napolitano M, Clipp E, Onken J, Farraye FA, Fletcher R. Prevalence and predictors of multiple behavioral risk factors for colon cancer. Prev Med. 2005 May;40(5):527-34. doi: 10.1016/j.ypmed.2004.10.001. PMID 15749134
- [Background] Prochaska JJ, Sallis JF. A randomized controlled trial of single versus multiple health behavior change: promoting physical activity and nutrition among adolescents. Health Psychol. 2004 May;23(3):314-8. doi: 10.1037/0278-6133.23.3.314. PMID 15099173
- [Background] Johnson SS, Paiva AL, Cummins CO, Johnson JL, Dyment SJ, Wright JA, Prochaska JO, Prochaska JM, Sherman K. Transtheoretical model-based multiple behavior intervention for weight management: effectiveness on a population basis. Prev Med. 2008 Mar;46(3):238-46. doi: 10.1016/j.ypmed.2007.09.010. Epub 2007 Oct 23. PMID 18055007
- [Background] Hyman DJ, Pavlik VN, Taylor WC, Goodrick GK, Moye L. Simultaneous vs sequential counseling for multiple behavior change. Arch Intern Med. 2007 Jun 11;167(11):1152-8. doi: 10.1001/archinte.167.11.1152. PMID 17563023
- [Background] Janz NK, Becker MH. The Health Belief Model: a decade later. Health Educ Q. 1984 Spring;11(1):1-47. doi: 10.1177/109019818401100101. PMID 6392204
- [Background] Becker MH. The Health Belief Model and personal health behavior. Becker MH, editor. San Francisco: Society for Public Health Education; 1974.
- [Background] Rosenstock IM, Strecher VJ, Becker MH. Social learning theory and the Health Belief Model. Health Educ Q. 1988 Summer;15(2):175-83. doi: 10.1177/109019818801500203. PMID 3378902
- [Background] Janz NK, Wren PA, Schottenfeld D, Guire KE. Colorectal cancer screening attitudes and behavior: a population-based study. Prev Med. 2003 Dec;37(6 Pt 1):627-34. doi: 10.1016/j.ypmed.2003.09.016. PMID 14636796
- [Background] Coleman EA, O'Sullivan P. Racial differences in breast cancer screening among women from 65 to 74 years of age: trends from 1987-1993 and barriers to screening. J Women Aging. 2001;13(3):23-39. doi: 10.1300/J074v13n03_03. PMID 11722004
- [Background] Green PM, Kelly BA. Colorectal cancer knowledge, perceptions, and behaviors in African Americans. Cancer Nurs. 2004 May-Jun;27(3):206-15; quiz 216-7. doi: 10.1097/00002820-200405000-00004. PMID 15238806
- [Background] Cooper GS, Koroukian SM. Racial disparities in the use of and indications for colorectal procedures in Medicare beneficiaries. Cancer. 2004 Jan 15;100(2):418-24. doi: 10.1002/cncr.20014. PMID 14716780
- [Background] Saywell RM Jr, Champion VL, Skinner CS, Menon U, Daggy J. A cost-effectiveness comparison of three tailored interventions to increase mammography screening. J Womens Health (Larchmt). 2004 Oct;13(8):909-18. doi: 10.1089/jwh.2004.13.909. PMID 15671706
- [Background] Champion V, Huster G. Effect of interventions on stage of mammography adoption. J Behav Med. 1995 Apr;18(2):169-87. doi: 10.1007/BF01857868. PMID 7563045
- [Background] Skinner CS, Arfken CL, Sykes RK. Knowledge, perceptions, and mammography stage of adoption among older urban women. Am J Prev Med. 1998 Jan;14(1):54-63. doi: 10.1016/s0749-3797(97)00008-1. PMID 9476836
- [Background] Champion VL, Skinner CS, Foster JL. The effects of standard care counseling or telephone/in-person counseling on beliefs, knowledge, and behavior related to mammography screening. Oncol Nurs Forum. 2000 Nov-Dec;27(10):1565-71. PMID 11103375
- [Background] Rakowski W, Fulton JP, Feldman JP. Women's decision making about mammography: a replication of the relationship between stages of adoption and decisional balance. Health Psychol. 1993 May;12(3):209-14. doi: 10.1037//0278-6133.12.3.209. PMID 8500450
- [Background] Rakowski W, Lefebvre RC, Assaf AR, Lasater TM, Carleton RA. Health practice correlates in three adult age groups: results from two community surveys. Public Health Rep. 1990 Sep-Oct;105(5):481-91. PMID 2120725
- [Background] Hovland CI, Janis IL, Kelley HH. Communication and Persuasion. Psychological studies of opinion change. New Haven: Yale University Press; 1953.
- [Background] Petty RE, Cacioppo JT. Attitudes and persuasion--classic and contemporary approaches. Boulder, CO: Westview Press; 1996.
- [Background] Champion V, Skinner CS, Menon U. Development of a self-efficacy scale for mammography. Res Nurs Health. 2005 Aug;28(4):329-36. doi: 10.1002/nur.20088. PMID 16028267
- [Background] Lairson DR, DiCarlo M, Myers RE, Wolf T, Cocroft J, Sifri R, Rosenthal M, Vernon SW, Wender R. Cost-effectiveness of targeted and tailored interventions on colorectal cancer screening use. Cancer. 2008 Feb 15;112(4):779-88. doi: 10.1002/cncr.23232. PMID 18098272
- [Background] Zapka JG, Lemon SC. Interventions for patients, providers, and health care organizations. Cancer. 2004 Sep 1;101(5 Suppl):1165-87. doi: 10.1002/cncr.20504. PMID 15329892
- [Background] Alexander GL, Divine GW, Couper MP, McClure JB, Stopponi MA, Fortman KK, Tolsma DD, Strecher VJ, Johnson CC. Effect of incentives and mailing features on online health program enrollment. Am J Prev Med. 2008 May;34(5):382-8. doi: 10.1016/j.amepre.2008.01.028. PMID 18407004
- [Background] Hall KL, Rossi JS. Meta-analytic examination of the strong and weak principles across 48 health behaviors. Prev Med. 2008 Mar;46(3):266-74. doi: 10.1016/j.ypmed.2007.11.006. Epub 2007 Nov 22. PMID 18242667
- [Background] Rakowski W, Dube CE, Marcus BH, Prochaska JO, Velicer WF, Abrams DB. Assessing elements of women's decisions about mammography. Health Psychol. 1992;11(2):111-8. doi: 10.1037//0278-6133.11.2.111. PMID 1582379
- [Background] Carlos RC, Fendrick AM, Patterson SK, Bernstein SJ. Associations in breast and colon cancer screening behavior in women. Acad Radiol. 2005 Apr;12(4):451-8. doi: 10.1016/j.acra.2004.12.024. PMID 15831418
- [Background] Morgan DL. Focus groups as qualitative research. 2nd ed. Thousand Oaks, CA: Sage Publications; 1997.
- [Background] Glaser BG, Strauss AL. The discovery of grounded theory: strategies for qualitative research. Paperback ed. Hawthorne, NY: Aldine de Gruyter; 1967.
- [Background] Lincoln YS, Guba EG. Naturalistic inquiry. Newbury Park: CA: Sage; 1985.
- [Background] Champion VL. Instrument development for health belief model constructs. ANS Adv Nurs Sci. 1984 Apr;6(3):73-85. doi: 10.1097/00012272-198404000-00011. PMID 6426380
- [Background] Champion VL. Revised susceptibility, benefits, and barriers scale for mammography screening. Res Nurs Health. 1999 Aug;22(4):341-8. doi: 10.1002/(sici)1098-240x(199908)22:43.0.co;2-p. PMID 10435551
- [Background] Champion VL. Instrument refinement for breast cancer screening behaviors. Nurs Res. 1993 May-Jun;42(3):139-43. PMID 8506161
- [Background] Rawl S, Champion VL, Menon U, Loehrer P, Vance G, Skinner CS. Validation of scales to measure benefits and barriers to colorectal cancer screening. Journal of Psychosocial Oncology. 2001;19(3/4):47-63.
- [Background] Kreuter MW, Strecher VJ. Changing inaccurate perceptions of health risk: results from a randomized trial. Health Psychol. 1995 Jan;14(1):56-63. doi: 10.1037//0278-6133.14.1.56. PMID 7737074
- [Background] Rawl S, Champion V, Menon U, Loehrer P, Vance G, Hunter C, et al. Differences on health beliefs by stage of readiness to screen for colorectal cancer among first-degree relatives of affected individuals. Ann Behav Med. 2001;23(Supplement):S202.
- [Background] Menon U. Factors associated with colorectal cancer screening in an average risk population [Dissertation]. Indianapolis, IN: Indiana University; 2000.
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Hosmer DW, Lemeshow S. Applied logistic regression. 2nd ed. New York: Wiley; 2000.
- [Background] Andersen MR, Hager M, Su C, Urban N. Analysis of the cost-effectiveness of mammography promotion by volunteers in rural communities. Health Educ Behav. 2002 Dec;29(6):755-70. doi: 10.1177/109019802237942. PMID 12456132
- [Background] Chirikos TN, Christman LK, Hunter S, Roetzheim RG. Cost-effectiveness of an intervention to increase cancer screening in primary care settings. Prev Med. 2004 Aug;39(2):230-8. doi: 10.1016/j.ypmed.2004.03.021. PMID 15226030
- [Background] Gold MR, Gold SR, Weinstein MC. Cost-effectiveness in health and medicine. Marthe R. Gold SRG, Milton C. Weinstein, editor. New York, NY: Oxford University Press; 1996.
- [Background] Drummond MF, Sculpher MJ, Torrance GW, O'Brien BJ, Stoddart GL. Methods for the economic evaluation of health care programmes. 3rd ed. Oxford: Oxford University Press; 2005.
- [Background] Briggs AH. Handling uncertainty in economic evaluation and presenting the results. Drummond M, Maguire, A., editor. Oxford: Oxford University Press; 2001.
- [Background] Westfall PH, Young SS. Resampling-based multiple testing: examples and methods for P-value adjustment. New York: Wiley; 1993.
- [Background] SPSS. Statistical package for the social sciences, 15.0 for Windows. 15.0 for Windows ed. Chicago: SPSS, Inc.; 2006.
- [Background] Dawson JD. Stratification of summary statistic tests according to missing data patterns. Stat Med. 1994 Sep 30;13(18):1853-63. doi: 10.1002/sim.4780131807. PMID 7997718
- [Derived] Huang D, Lairson DR, Chung TH, Monahan PO, Rawl SM, Champion VL. Economic Evaluation of Web- versus Telephone-based Interventions to Simultaneously Increase Colorectal and Breast Cancer Screening Among Women. Cancer Prev Res (Phila). 2021 Sep;14(9):905-916. doi: 10.1158/1940-6207.CAPR-21-0009. Epub 2021 Jul 9. PMID 34244154
- [Derived] Champion VL, Christy SM, Rakowski W, Lairson DR, Monahan PO, Gathirua-Mwangi WG, Stump TE, Biederman EB, Kettler CD, Rawl SM. An RCT to Increase Breast and Colorectal Cancer Screening. Am J Prev Med. 2020 Aug;59(2):e69-e78. doi: 10.1016/j.amepre.2020.03.008. PMID 32690203
- [Derived] Lairson DR, Chung TH, Huang D, Stump TE, Monahan PO, Christy SM, Rawl SM, Champion VL. Economic Evaluation of Tailored Web versus Tailored Telephone-Based Interventions to Increase Colorectal Cancer Screening among Women. Cancer Prev Res (Phila). 2020 Mar;13(3):309-316. doi: 10.1158/1940-6207.CAPR-19-0376. Epub 2020 Jan 22. PMID 31969343

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2014-01-24): https://cdn.clinicaltrials.gov/large-docs/98/NCT03279198/Prot_SAP_000.pdf
  • Informed Consent Form (2014-06-11): https://cdn.clinicaltrials.gov/large-docs/98/NCT03279198/ICF_001.pdf